CLINICAL TRIAL: NCT06054399
Title: Education Project on Migraine in Pregnant Women Attended at Clínica Alemana de Santiago, Chile
Brief Title: Education on Migraine in Pregnant Women
Acronym: MIGREMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, Veronica Olavarria, Medical Doctor, Clinica Alemana de Santiago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MIGREMB Study
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Migraine Disorders
Keywords: migraine; pregnancy
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: before and after quasi experimental
Masking Description: All the participants will know about the educational interventional as well as their physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Audiovisual educational intervention (Experimental): Audiovisual educational intervention will be apply within 3 moments of the pregnancy pf patients.
  Interventions: Other: educational program

INTERVENTIONS:
Other: educational program — Education resources in Spanish through social media directed to the targeted audience mentioned above. There will be at least three interventions along the study, one for each pregnancy trimester, including topics such as: Migraine criteria, management strategies, risks of medication overuse, alarm symptoms, etc. These educational interventions will be conducted by trained health care professionals, mainly using audio-visual media.

SUMMARY:
Patient education is one type of low-cost intervention that can be easily applied but there are not specific studies about it in pregnant women with migraine.

The primary goal of the study is to educate pregnant women experiencing migraine, leading to their understanding of the underlying pathology, management strategies and alarm symptoms.

An intervention based on education can lead to empowered individuals capable of self-management, therefore reducing medication overuse and inappropriate use of the emergency department.

It is relevant that these patients have access to understandable information; that is, in their own language and avoiding complex medical terms, so that the information can be useful for them and their support system.

With this project the investigators aimed to improve the knowledge and satisfaction of participants (patients and healthcare professionals) to better deal with migraines during pregnancy.

DETAILED DESCRIPTION:
The primary aim of the study is to educate pregnant women experiencing migraine, leading to their understanding of the underlying pathology, management strategies and alarm symptoms.

The target population are pregnant women suffering from migraine in prenatal follow-up in Clínica Alemana (Santiago, Chile). Included as a secondary target population are the obstetricians following these patients. The investigators propose to design an educational intervention. The investigators will develop education material about migraine in Spanish and the study team will work using social media and some basic material on paper. The investigators will educate first obstetricians of the institution (Clínica Alemana de Santiago) and will work with the obstetricians in the recruitment of patients (according to International Classification of Headache Diseases-3 (ICHD-3) criteria. Secondly, among patients who consent, three educational interventions will be apply along their pregnancy, considering topics like the knowledge of migraine criteria, management strategies and alarm symptoms.

In this project two scores will be measured in pregnant women, both at their first prenatal appointment and at the end of their postpartum period (up to 42 days postpartum). These are: Migraine Disability Assessment questionnaire, and the Brief Illness Perception questionnaire, to evaluate cognitive and emotional representation of illness. Among obstetricians, the investigators will prepare and deliver a short questionnaire with dichotomous questions to evaluate their sense of knowledge regarding migraine, the satisfaction with the study and the importance the obstetricians give to the newly acquired information on daily practice.

The project will last 2 years in total, of which patients will be recruited for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years or older with migraine according to clinical criteria
* Informed Consent signed
* Controlled during its pregnancy at Clínica Alemana de Santiago

Exclusion Criteria:

* Any impossibility to complete the follow-up during postpartum period.
* Language barriers that would impede the patient to understand the applied questionnaires and educational interventions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Migraine Disability Assessment questionnaire score | 8 to 9 months
  The Migraine Disability Assessment questionnaire will be apply to patients, both at their first prenatal appointment and at the end of their postpartum period (up to 42 days postpartum), to evaluate the level of pain and the impact of headache on their daily life.The questionnaire comprises 7 questions in total and the score ranges between 0 to 90, higher scores mean higher grade of disability.
Improvement in Brief Illness Perception questionnaire score | 8 to 9 months
  Both at their first prenatal appointment and at the end of their postpartum period (up to 42 days postpartum), the Brief Illness Perception questionnaire, to evaluate cognitive and emotional representation of illness.This questionnaire comprises 8 items and the score ranges from 0 to 80, a higher score indicates a greater perceived psychological burden of illness.

SECONDARY OUTCOMES:
Obstetricians Assessment | 9 months
  A survey will be delivered with dichotomous questions to evaluate their sense of knowledge regarding migraine, their satisfaction with the study and the importance they give to the newly acquired information on their daily practice.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica V Olavarria, MD, MSC, Principal Investigator — Clinica Alemana de Santiago
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No